CLINICAL TRIAL: NCT04373057
Title: A Phase I/II Trial of the Prebiotic Galacto-oligosaccharide to Prevent Acute GVHD
Brief Title: Prebiotic Galacto-oligosaccharide and Acute GVHD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00105137
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Acute GVHD
MeSH Terms: interventions — 4'-galactooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galacto-oligosaccharide (Experimental): Phase I: Subjects will receive GOS, at dose levels 0.75g, 1.5g, and 2.9 g/day administered once daily. GOS will be dosed per the following schedule using a modified 3+3 design: 0.75g x 4 days, followed by 1.5g x 4 days, followed by 2.9g for the duration of the study starting from about 30 days before transplant to about 4 weeks after transplant.
  Phase II: Subjects will receive GOS, at dose levels 0.25*MTD, 0.5*MTD, and MTD with MTD determined by the phase 1 of the study, once daily from about 30 days before transplant to about 4 weeks after transplant.
  Interventions: Dietary Supplement: Galacto-oligosaccharide
- Maltodextrin (Placebo Comparator): Phase II: Subjects will receive maltodextrin at comparable dose level as GOS (in Phase II) once daily from about 30 days before transplant to about 4 weeks after transplant.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharide — GOS will be administered at determined dose levels per protocol once daily from about 30 days before transplant to about 4 weeks after transplant.
  Other Names: Bimuno®, B-GOS
  Arms: Galacto-oligosaccharide
Dietary Supplement: Maltodextrin — Maltodextrin will be administered at comparable dose level as GOS (in Phase II) once daily from about 30 days before transplant to about 4 weeks after transplant.
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to determine whether the carbohydrate prebiotic (dietary supplement) known as galacto-oligosaccharide (GOS) can modulate the microbiome (the bacteria in the gut) and help prevent graft-versus host disease (GVHD) after allogeneic stem cell transplant. The study has two two parts. In phase 1, the best dose of GOS will be evaluated. In phase 2, using the best dose of GOS, participants will be randomized to receive GOS or a placebo (maltodextrin, a common food additive that is not known to affect the microbiome) so that the effect of GOS can be determined.

DETAILED DESCRIPTION:
Humans carry on the order of 100 trillion microbial cells (the microbiota),which play a major role in normal health as well as disease pathogenesis. In the gut, the microbiota interact with the intestinal epithelium and immune system to regulate inflammation and metabolism. The impact of the microbiota on GVHD and other clinical outcomes may be mediated by bacterial metabolites such as short chain fatty acid (SCFAs). In particular, the SCFA butyrate has been shown to be a preferred fuel source of human colonic epithelial cells and essential for normal differentiation of regulatory immune cells in the intestine, which in turn may decrease GVHD. This is supported by murine studies, in which manipulating the gut microbiota to increase microbial SCFA production or by direct administration (oral gavage) of butyrate has been shown to improve HCT outcomes, including protection from GVHD

Manipulating the gut microbiota in HCT to decrease the risk of GVHD could potentially be done using several methods, namely prebiotics (dietary carbohydrates or fibers), probiotics (live bacteria), and fecal transplantation. In contrast to live bacteria, prebiotics are dietary carbohydrates classified as nutritional supplements that can sustain gut bacteria, regulate gastrointestinal transit time, and foster cooperative metabolic networks between enteric microbes. Because prebiotics encourage the growth of existing bacteria rather than introducing new organisms, they may be safer. Moreover, bacterial fermentation of prebiotics may yield SCFA.

The purpose of this study is to determine whether the carbohydrate prebiotic (dietary supplement) known as galacto-oligosaccharide (GOS) can modulate the microbiome (the bacteria in the gut) and help prevent graft-versus host disease (GVHD) after allogeneic stem cell transplant. The study has two two parts. In phase 1, three dose levels 0.75g/day (25% maximum dose, D1), 1.5g/day (50% maximum dose D2), and 2.9g/day (maximum dose, D3) will be evaluated to find out the provisional maximum tolerated dose (pMTD) of GOS to be used in phase 2. In phase 2, using pMTD of GOS, participants will be randomized to receive GOS or a placebo (maltodextrin, a common food additive that is not known to affect the microbiome) so that the effect of GOS can be determined. Note that if the pMTD is D3, there will be a D1 and D2 lead-in period similar to the Phase 1 study however if the pMTD is D2, there will only be a lead-in with D1 and if pMTD is D1, there will only be one dose with no lead-in. The study will generate important data on gut microbiota responses to help tailor or personalize future prebiotic therapies to patients and their microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Plan to undergo allogeneic HCT for any cancer or non-cancer illness
* Age 18-80 years
* Karnofsky Performance Status >70

Exclusion Criteria:

* Pregnant/lactating
* Malabsorption syndrome, short bowel or chologenic diarrhea
* At time of enrollment, Grade 2 or higher GI symptoms per NCI-CTCAE
* Active treatment with other prebiotics, probiotics, or herbal supplementation (ok if stops before enrollment)
* Active treatment with antibiotics (with the exception of prophylactic antibiotics)
* Concurrent enrollment on the Duke HCT Home Transplant study or another clinical trial targeting GVHD; patients who are enrolled in observational or non-pharmacologic intervention trials (for example, the Duke HCT Research-POP Pre and Peri-HCT Optimization Program aka "R-POP") or pharmacologic or cellular therapy trials with other targets (for example, NK DLI) are NOT excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
provisional Maximum Tolerated Dose (pMTD) of GOS | 30 days
  GOS will be dosed as outlined using a modified 3+3 design: 0.75g x 4 days, followed by 1.5g x 4 days, followed by 2.9g for the duration of the study. If two or more subjects experience new grade 2 or 3 pre-HCT toxicities at a given dose level, that dose will be considered not tolerable and the previous dose pMTD. If two or more subjects experience new grade 2 or higher pre-HCT toxicities at the 0.75g/day dose, study may be paused to revisit the design. If one subject experiences new grade 2 or 3 pre-HCT toxicities at a given dose level, additional 3 subjects will be enrolled at this same dose schedule. If one or more of these additional subjects experience new grade 2 or 3 pre-HCT toxicities at that same or lower dose level, this dose level will be considered not tolerable and the previous dose the pMTD. If no subjects experience new grade 2 or 3 pre-HCT toxicities or only one of six subjects experience new grade 2 or 3 pre-HCT toxicities, 2.9g/day dose will be assumed to be the pMTD
Incidence of Grade II-IV acute GVHD at Day 100 | 100 days
  Acute GVHD Scoring will be done following BMT CTN, 2013 criteria.

SECONDARY OUTCOMES:
Incidence of acute GI toxicities through Day 30 | 30 days
  Acute GI toxicities include mucositis, nausea, vomiting, diarrhea, constipation, abdominal pain, and bloating through D30 as assessed by CTCAE v5.
Incidences of Acute GI toxicities as measured by self-reported evaluation through Day 30 | 30 days
  Acute GI toxicities as measured by self-reported (PRO-CTCAE) evaluation of decreased appetite, anxiety, sadness, fatigue, insomnia, general pain, shortness of breath, numbness and tingling, mouth sores, nausea, vomiting, diarrhea, constipation, abdominal pain, and bloating through D 30 (5 point ordinal scale per PRO-CTCAE)
Incidence of chronic GVHD at Day 365 and Day 730 | Day 365 and day 730
  Chronic GVHD Scoring will be done following NIH Consensus Criteria
Health care utilization through Day 100, through Day 365, and through Day 730 | Day 100, Day 365, and Day 730
  Data will be obtained through chart review at or after Day 100, Day 365, and Day730 (respectively), and will be reported as means/medians depending on the distribution of data (for example, mean/median health care utilization through Day 100)
Overall survival (OS) at Day 365 and Day 730 | Day 365 and Day 730
  Data will be obtained by chart review at or after D365 and D730 Data will be reported as a percentage (ie. 1-year and 2-year overall survival) for each arm
Relapse-free survival (RFS) at Day 365 and Day 730 | Day 365 and Day 730
  Data will be obtained by chart review at or after Day 365 and Day 730 Data will be reported as a percentage (ie. 1-year and 2-year overall survival) for each arm
Total parenteral nutrition (TPN) use through Day 30 and Day 100 | Day 30 and Day 100
  Data will be obtained as part of the GVHD Prophylaxis/medication assessments. Data will be reported as a percentage for each arm (at each of the time points)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke Health; Anthony Sung, MD, Principal Investigator — University of Kansas
Locations (2):
- United States (2):
  - Kansas University Medical Center, Kansas City, Kansas
  - Duke, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lakshmanan AP, Deola S, Terranegra A. The Promise of Precision Nutrition for Modulation of the Gut Microbiota as a Novel Therapeutic Approach to Acute Graft-versus-host Disease. Transplantation. 2023 Dec 1;107(12):2497-2509. doi: 10.1097/TP.0000000000004629. Epub 2023 May 16. PMID 37189240